CLINICAL TRIAL: NCT02648308
Title: Extension of the 5As Team Study for Improved Provider Obesity Management to Physicians and Medical Trainees (Part 2)
Acronym: 5AsT-MD2
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other)
Responsible Party: Principal Investigator, Denise Campbell, Associate Professor, Department of Family Medicine, University of Alberta, University of Alberta
Other Study IDs: Pro00058323
Record Dates: First submitted 2015-10-21; First posted 2016-01-07 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Obesity
Keywords: Education, Medical
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Obesity Management Workshop — Workshop provided to first year medical residents to improve confidence and skill when conducting weight management visits with patients

SUMMARY:
Results from the 5As Team (5AsT) Study have identified critical gaps in medical school curricula on obesity, leading to a wave of new family physicians who lack confidence and are poorly equipped to manage obesity with their patients. In an effort to address this gap, all first year medical residents training in family medicine at the University of Alberta during the 2015/2016 year will be required to take a 2 day workshop in Obesity Management as part of the Doctor-Patient Relationship Course. The comprehensive workshop provides medical residents with knowledge and training in obesity prevention and management through didactic lectures, experiential learning, and clinical practice. Participants were asked to complete and submit pre- and post- workshop assessment measuring self-reported confidence on aspects of weight management counselling, narrative reflections regarding the experiential components of the course, and measures to assess beliefs and attitudes towards people living with obesity. The purpose of our program evaluation was to assess the program's impact on residents' knowledge of obesity and attitude towards counselling patients with obesity, as well as to refine and further develop the course. Evaluation of the 5AsT-MD pilot project shows increases of residents' understanding of the complexity and chronicity of obesity, and an uptake of the 5As framework and tools by residents to improve confidence and success of their weight management practice.

DETAILED DESCRIPTION:
Background:

Obesity is a complex chronic condition that negatively impacts individuals, society, and the healthcare system. Family physicians are one of many health practitioners tasked with the long-term care of patients with obesity and its associated co-morbidities. However, focus groups conducted by the 5As Team (5AsT) have identified critical gaps in medical school curricula on obesity, leading to a wave of new family physicians who are unconfident and poorly equipped to manage obesity with their patients. To address this education gap, the 5As team developed a comprehensive training module on obesity management for family medicine residents at the University of Alberta.

Study Objectives:

This study aimed to evaluate the impact of this course on the residents' attitudes and beliefs about obesity, as well as confidence levels using key aspects of the 5As of obesity management to help their patients.

Methods:

Based on focus groups conducted with medical students and practicing physicians during a summer project, a list of learning objectives was made to address known deficiencies in obesity education. These learning objectives were adapted to a two-day training module on obesity management for first year family medicine residents. All 2015/2016 and 2016/2017 first year medical residents were required to take a 2 day Obesity Management Workshop as part of their Doctor-Patient Relationship course. Prior to the workshop, residents were asked to complete a pre-workshop assessment which asked them to rate their level of confidence counselling patients on several aspects of obesity management. In addition, residents enrolled in the year 2015/2016 were asked to complete the Attitudes Toward Obese Persons (ATOP) and Beliefs About Obese Persons BAOP questionnaires, residents enrolled in the 2016/2017 year were asked to complete the NEW Attitudes Scale. The first day consisted of didactic lectures on the basic pathophysiology of obesity, obesity management in pediatrics and pregnancy, and an introduction to the 5As of obesity management. Residents were also given the opportunity to experience wearing a bariatric suit in a simulated living environment after which they were asked to complete their first narrative reflection assignment. The second day of the workshop consisted of didactic lectures on lifestyle management and bariatric surgery, followed by practice sessions with standardized patients. Residents were then asked to find a patient with lived experience in their own clinic and practice using the 5As approach with their own patient and then complete their second narrative reflection assignment.

Consent:

Residents were informed about the 5AsT MD2 study on the first day of the 2-day workshop and asked if they would like to participate. If a resident declined to participate, they were still able to take part in the workshop and were still required to complete the course assignments listed above, however, their course materials were not provided to the research team.

Study Procedures:

Those residents who consented to participate in the study, were asked to place their required course materials into a sealed envelope and will then submit them to a neutral, third party. The neutral, third party was an employee in the Department of Family Medicine and had no responsibilities with regards to evaluation of the medical residents. The neutral, third party recorded that the resident had completed their assignment for the course, assigned an Identification (ID) number to each resident and labelled each document as well as the envelope with the resident's ID number. Using a paper cutter, the neutral, third party removed the resident's name from each document. A master list was kept by the neutral, third party, which allowed her to track which ID number corresponded to which resident so that she could appropriately label all of the post-workshop documents with the resident's assigned ID number. Only the neutral, third party had access to the master last with the residents names.

Following the workshop on the second day, the residents who consented to participate, were asked to submit their post-workshop course materials, in a sealed envelope, to the neutral third party. The neutral, third party recorded that the resident completed their assignment for the course, labelled their documents and envelope with the correct ID number and then removed the resident's name from the documents. The de-identified materials of those residents who consented to participate were given to study staff. The narrative reflective exercises for both part 1 and part 2 of the workshop were due 2 weeks post-workshop event.

Results:

Participants completed the validated ATOP (Attitudes Toward Obese Persons) and BAOP (Beliefs About Obese Persons) questionnaires, as well as pre- and post- workshop assessment questionnaires to measure their level of confidence in performing key aspects of obesity management. All questionnaires were de-identified, but responses were tracked both before and after the training module to quantify the change seen in each study participant. Participants also wrote two de-identified narrative reflections to be used for qualitative analysis. The first was on the weight bias bariatric suit experience, and the second was on the application of the lessons of the workshop in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be first year medical residents training in family medicine at the University of Alberta. They will be recruited from the Obesity Management Workshop that is a required component of their course on Doctor-Patient Relationships. All participants must be over the age of 18 and be able to communicate effectively in English.

Exclusion Criteria:

* If participants are unable to communicate effectively in English, they will not be able to participate in the study. The Obesity Management Workshop will be presented in English and participants must be able to understand the presentation and written documents that they are being asked to complete.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: First year medical residents who are training in family medicine at the University of Alberta.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2015-10-08 (Actual); Primary Completion 2017-04-06 (Actual); Study Completion 2017-08-27 (Actual)

PRIMARY OUTCOMES:
Changes in Attitudes Towards Obese Persons (ATOP) | baseline, 3 weeks
  Self-reported measure about a person's attitudes towards obese persons to see whether their attitude towards people living with obesity changed as a result of the knowledge gained through the obesity management workshop.
Changes in Beliefs About Obese Persons (BAOP) | baseline, 3 weeks
  Self-reported measure about a person's beliefs about obese persons to see whether their beliefs about people living with obesity changed as a result of the knowledge gained through the obesity management workshop.
Changes in Self-Reported Comfort Level (Pre- and Post- Assessment Scale) | baseline, 3 weeks
  The pre- and post- questionnaire is a self-reported measure of the resident's comfort level around each of the 5 areas of the 5A's Obesity Management. Questions related to each element of the 5A's are rated using a 5 point Likert Scale.
Qualitative: Narrative Reflections | baseline, 3 weeks
  Personal reflection on how the experience and the workshop made the person feel. These will be analyzed using qualitative analysis to see how the workshop may have affected views, beliefs and their practice.

CONTACTS AND LOCATIONS:
Overall Officials: Denise L Campbell-Scherer, MD, PhD, Principal Investigator — University of Alberta, Department of Family Medicine; Arya Sharma, Principal Investigator — University of Alberta, Faculty of Medicine
Locations (1):
- University of Alberta - Department of Family Medicine, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Asselin J, Osunlana AM, Ogunleye AA, Sharma AM, Campbell-Scherer D. Missing an opportunity: the embedded nature of weight management in primary care. Clin Obes. 2015 Dec;5(6):325-32. doi: 10.1111/cob.12115. Epub 2015 Aug 25. PMID 26303812
- [Background] Osunlana AM, Asselin J, Anderson R, Ogunleye AA, Cave A, Sharma AM, Campbell-Scherer DL. 5As Team obesity intervention in primary care: development and evaluation of shared decision-making weight management tools. Clin Obes. 2015 Aug;5(4):219-25. doi: 10.1111/cob.12105. Epub 2015 Jun 30. PMID 26129630
- [Background] Campbell-Scherer DL, Asselin J, Osunlana AM, Fielding S, Anderson R, Rueda-Clausen CF, Johnson JA, Ogunleye AA, Cave A, Manca D, Sharma AM. Implementation and evaluation of the 5As framework of obesity management in primary care: design of the 5As Team (5AsT) randomized control trial. Implement Sci. 2014 Jun 19;9:78. doi: 10.1186/1748-5908-9-78. PMID 24947045